CLINICAL TRIAL: NCT07216898
Title: You Have the Right to Know: Empowering Women Through Clean Beauty Research and Education
Brief Title: Clean Beauty in Newark, NJ
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Emily S. Barrett, PhD, Vice Chair, Department of Biostatistics and Epidemiology, Rutgers, The State University of New Jersey
Other Study IDs: Pro2025001147; P30ES005022 (NIH)
Record Dates: First submitted 2025-10-03; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Health Disparities; Education
Keywords: Endocrine Disrupting Chemicals; Personal Care Products; Environmental Health Disparities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Clean Beauty Event Attendees: Participants in clean beauty events will be educated on the risks of toxic chemicals in personal care products and safer alternatives. They will be invited to provide information on their personal care product use and buying habits immediately before and after the educational events. Three months after the events, participants will complete surveys on any sustained changes in product use behaviors.
  Interventions: Behavioral: Chemical Exposure Prevention

INTERVENTIONS:
Behavioral: Chemical Exposure Prevention — Education on potential toxic chemicals found within personal care products and safer alternatives during community-engaged clean beauty events.

SUMMARY:
Every day, consumers use personal care products containing thousands of manmade chemicals. Growing evidence suggests that personal care products specifically marketed to Black women (e.g., hair straighteners and oils, skin lighteners) often contain potentially hazardous chemicals that can interfere with hormones or increase cancer risks. This research focuses on how the investigators can educate and activate community members in Newark, NJ to reduce disparities in exposures occurring through hair products. Leveraging educational clean beauty events hosted by collaborators at Clean Water Action, the investigators will administer surveys on hair product use and attitudes immediately before and after a clean beauty educational intervention. Participants will also complete surveys 3 months post-event to examine any changes in attitudes or behaviors around hair products and their use and safety.

DETAILED DESCRIPTION:
The investigators will evaluate hair product perceptions, knowledge, and use among community members before and after an educational intervention. At the beginning of Clean Beauty events hosted by Clean Water Action, the investigators will collect survey data on hair product use as well as knowledge and perceptions around product safety from attendees. The investigators will administer a post-workshop survey to evaluate changes in knowledge and perceptions from pre- to post-workshop. Three months after the workshop, the investigators will distribute a follow-up survey to examine whether the intervention had sustained impacts on hair product perceptions, knowledge, or use.

ELIGIBILITY:
Inclusion Criteria:

* Attendees of clean beauty events hosted by Clean Water Action, age 18 and older

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Attendees of clean beauty events hosted by Clean Water Action
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is any intended changes in participants' hair routines from pre to post event | The outcome will be assessed immediately post-event (1-2 hours after baseline).
  After the Clean Beauty intervention event, participants will be asked, "Based on what you learned today, do you think you will make any changes to your hair style, hair routine, or the products you use?" [Answer choices: Yes/No/Not sure] We will calculate the percentage of participants who plan to make a change in their hair routine.

SECONDARY OUTCOMES:
Perceptions of hair product safety following the Clean Beauty intervention event. | Changes in perceptions around hair product safety will be evaluated 3 Months after baseline.
  Our main secondary outcome is changes in perceptions around hair product safety from before the Clean Beauty intervention event to three months after the event. Prior to the event, at baseline, participants will be asked the extent to which they agree with the statement that "The hair products I use affect my health" (Answer choices: Strongly disagree, disagree, neither agree nor disagree, agree, strongly agree). The question will be repeated in a three month follow-up questionnaire. We will look at changes from baseline to the three month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Barrett, PhD, Principal Investigator — Rutgers School of Public Health
Locations (1):
- Weequahic Park, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
The results of this study are only relevant to scientific knowledge when considered on an aggregate level.

REFERENCES:
- [Background] Wright MA, Moore KR, Upson K, Baird DD, Chin HB. Douching or Perineal Talc Use and Prevalent Fibroids in Young African American Women. J Womens Health (Larchmt). 2021 Dec;30(12):1729-1735. doi: 10.1089/jwh.2020.8524. Epub 2021 Mar 5. PMID 33667128
- [Background] White AJ, Sandler DP, Gaston SA, Jackson CL, O'Brien KM. Use of hair products in relation to ovarian cancer risk. Carcinogenesis. 2021 Oct 5;42(9):1189-1195. doi: 10.1093/carcin/bgab056. PMID 34173819
- [Background] Silbergeld EK, Mandrioli D, Cranor CF. Regulating chemicals: law, science, and the unbearable burdens of regulation. Annu Rev Public Health. 2015 Mar 18;36:175-91. doi: 10.1146/annurev-publhealth-031914-122654. PMID 25785889
- [Background] Johnson PI, Favela K, Jarin J, Le AM, Clark PY, Fu L, Gillis AD, Morga N, Nguyen C, Harley KG. Chemicals of concern in personal care products used by women of color in three communities of California. J Expo Sci Environ Epidemiol. 2022 Nov;32(6):864-876. doi: 10.1038/s41370-022-00485-y. Epub 2022 Nov 2. PMID 36323919
- [Background] Zota AR, Shamasunder B. The environmental injustice of beauty: framing chemical exposures from beauty products as a health disparities concern. Am J Obstet Gynecol. 2017 Oct;217(4):418.e1-418.e6. doi: 10.1016/j.ajog.2017.07.020. Epub 2017 Aug 16. PMID 28822238
- [Background] James-Todd TM, Chiu YH, Zota AR. Racial/ethnic disparities in environmental endocrine disrupting chemicals and women's reproductive health outcomes: epidemiological examples across the life course. Curr Epidemiol Rep. 2016 Jun;3(2):161-180. doi: 10.1007/s40471-016-0073-9. Epub 2016 Mar 31. PMID 28497013
- [Background] Preston EV, Chan M, Nozhenko K, Bellavia A, Grenon MC, Cantonwine DE, McElrath TF, James-Todd T. Socioeconomic and racial/ethnic differences in use of endocrine-disrupting chemical-associated personal care product categories among pregnant women. Environ Res. 2021 Jul;198:111212. doi: 10.1016/j.envres.2021.111212. Epub 2021 May 3. PMID 33957140
- [Background] Welch BM, Keil AP, Buckley JP, Engel SM, James-Todd T, Zota AR, Alshawabkeh AN, Barrett ES, Bloom MS, Bush NR, Cordero JF, Dabelea D, Eskenazi B, Lanphear BP, Padmanabhan V, Sathyanarayana S, Swan SH, Aalborg J, Baird DD, Binder AM, Bradman A, Braun JM, Calafat AM, Cantonwine DE, Christenbury KE, Factor-Litvak P, Harley KG, Hauser R, Herbstman JB, Hertz-Picciotto I, Holland N, Jukic AMZ, McElrath TF, Meeker JD, Messerlian C, Michels KB, Newman RB, Nguyen RHN, O'Brien KM, Rauh VA, Redmon B, Rich DQ, Rosen EM, Schmidt RJ, Sparks AE, Starling AP, Wang C, Watkins DJ, Weinberg CR, Weinberger B, Wenzel AG, Wilcox AJ, Yolton K, Zhang Y, Ferguson KK. Racial and Ethnic Disparities in Phthalate Exposure and Preterm Birth: A Pooled Study of Sixteen U.S. Cohorts. Environ Health Perspect. 2023 Dec;131(12):127015. doi: 10.1289/EHP12831. Epub 2023 Dec 20. PMID 38117586
- [Background] Manuck TA. Racial and ethnic differences in preterm birth: A complex, multifactorial problem. Semin Perinatol. 2017 Dec;41(8):511-518. doi: 10.1053/j.semperi.2017.08.010. Epub 2017 Sep 21. PMID 28941962
- [Background] Giaquinto AN, Sung H, Newman LA, Freedman RA, Smith RA, Star J, Jemal A, Siegel RL. Breast cancer statistics 2024. CA Cancer J Clin. 2024 Nov-Dec;74(6):477-495. doi: 10.3322/caac.21863. Epub 2024 Oct 1. PMID 39352042
- [Background] Katon JG, Plowden TC, Marsh EE. Racial disparities in uterine fibroids and endometriosis: a systematic review and application of social, structural, and political context. Fertil Steril. 2023 Mar;119(3):355-363. doi: 10.1016/j.fertnstert.2023.01.022. Epub 2023 Jan 20. PMID 36682686
- [Background] Llanos AAM, Rockson A, Getz K, Greenberg P, Portillo E, McDonald JA, Teteh DK, Villasenor J, Lozada C, Franklin J, More V, Rivera-Nunez Z, Kinkade CW, Barrett ES. Assessment of personal care product use and perceptions of use in a sample of US adults affiliated with a university in the Northeast. Environ Res. 2023 Nov 1;236(Pt 1):116719. doi: 10.1016/j.envres.2023.116719. Epub 2023 Jul 21. PMID 37481059
- [Background] Payne CE, Rockson A, Ashrafi A, McDonald JA, Bethea TN, Barrett ES, Llanos AAM. Beauty Beware: Associations between Perceptions of Harm and Safer Hair-Product-Purchasing Behaviors in a Cross-Sectional Study of Adults Affiliated with a University in the Northeast. Int J Environ Res Public Health. 2023 Nov 30;20(23):7129. doi: 10.3390/ijerph20237129. PMID 38063560